CLINICAL TRIAL: NCT01938755
Title: Hyperbaric Levobupivacaine for Spinal Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, özgür yağan, Özgür Yağan, Ordu University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: odu52
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: This Study Was Focused on Selective Spinal Anesthesia for Lower Extremity Surgery in Order to Achieve Early Mobilization and to Shorten Hospital Stay
MeSH Terms: interventions — Levobupivacaine

ARMS (3):
- levobupivacaine I (Experimental): group that was administered levobupivacaine plus 60mg dextrose
  Interventions: Drug: levobupivacaine
- levobupivacaine II (Experimental): group that was administered levobupivacaine plus 80 mg dextrose
  Interventions: Drug: levobupivacaine
- levobupivacaine III (Experimental): group that was administered levobupivacaine plus 100 mg dextrose
  Interventions: Drug: levobupivacaine

INTERVENTIONS:
Drug: levobupivacaine — levobupivacaine plus 60 mg dextrose
  Arms: levobupivacaine I
Drug: levobupivacaine — levobupivacaine plus 80 mg dextrose
  Arms: levobupivacaine II
Drug: levobupivacaine — levobupivacaine plus 100 mg dextrose
  Arms: levobupivacaine III

SUMMARY:
Spinal anaesthesia also called spinal block or sub-arachnoid block (SAB), is a form of regional anaesthesia involving injection of a local anaesthetic into the subarachnoid space, generally through a fine needle.

There is no generic hyperbaric form of levobupivacaine currently available so we aimed in this study that to find the appropriate concentration of the levobupivacaine which achieves unilateral spinal anesthesia. The potential benefits of this type of anesthesia are less motor blockade and urinary retention, decrease in hospital stay. Therefore, it seems to be suitable for outpatient anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Approval to participate in the study and spinal anesthesia
* American society of anesthesia (ASA) I,II physical status
* Scheduled for lower extremity surgery

Exclusion Criteria:

* Refuse to participate in the study
* American society of anesthesia (ASA)III, IV physical status
* Hypersensitivity to local anesthetics
* Emergency surgery
* Chronic pain treatment
* Peripheral neuropathy
* Severe systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
degree of motor blockade | until dissolve of motor blockade

CONTACTS AND LOCATIONS:
Locations (1):
- Anestesia and Reanimation Dept.; Ordu University Education and Research Hospital, Ordu, Ordu, Turkey (Türkiye)